CLINICAL TRIAL: NCT00001249
Title: Treatment of Tac-Expressing Cutaneous T-Cell Lymphoma (CTCL) and Adult T-Cell Leukemia (ATL) With Yttrium-90 Radiolabeled Anti-Tac
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 900043; 90-C-0043
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-11

CONDITIONS: Leukemia, T-Cell; Lymphoma, T-Cell, Cutaneous
Keywords: Interleukin-2 Receptor
MeSH Terms: conditions — Leukemia, T-Cell; Lymphoma, T-Cell, Cutaneous; Diabetes Mellitus, Insulin-Dependent, 10

INTERVENTIONS:
Drug: Yttrium-90 radiolabeled anti-Tac antibody

SUMMARY:
The study purpose is to evaluate the clinical response to multidose administration of anti-Tac monoclonal antibody conjugated with 10 mCi 90Y in patients with Tac-expressing adult T-cell leukemia (ATL).

DETAILED DESCRIPTION:
The study purpose is to evaluate the clinical response to multidose administration of anti-Tac monoclonal antibody conjugated with 10 mCi 90Y in patients with Tac-expressing adult T-cell leukemia (ATL). This study represents an extension of phase I trial (Clinical Project #90-C-0043, FDA IND #3469) which permitted the administration of 5 mCi, 10 mCi, and 15mCi 90Y-anti-Tac to patients with ATL. We propose to administer 90Y-anti-Tac (10 mCi doses) to patients with Tac-expressing ATL who are over 18 years of age and who fill the patient eligibility criteria.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Histologically confirmed adult T-cell leukemia/lymphoma (ATL) or cutaneous T-cell lymphoma (CTCL).

Reactivity of at least 10% of peripheral blood, lymph node, or dermal malignant cells with anti-Tac as determined by immunofluorescent staining or soluble IL-2 receptor level greater than 1,500 U required.

All stages of Tac-expressing T-cell leukemia and lymphoma eligible except Stage I CTCL.

All forms of ATL eligible, including the "smoldering" type as well as aggressive disease.

No symptomatic CNS disease other than tropical spastic paraparesis.

Asymptomatic CNS disease with demonstrable malignant cells in the CSF allowed (such patients receive CNS therapy, e.g., intrathecal methotrexate and/or CNS irradiation, as appropriate).

PRIOR/CONCURRENT THERAPY:

Biologic Therapy: Not specified.

Chemotherapy:

CTCL must have failed initial chemotherapy.

ATL may or may not have had prior chemotherapy.

At least 4 weeks since prior cytotoxic chemotherapy.

Endocrine Therapy: Not specified.

Radiotherapy: At least 4 weeks since prior radiotherapy.

Surgery: Not specified.

PATIENT CHARACTERISTICS:

Age: 18 and over.

Performance status: Not specified.

Life expectancy: Greater than 1 month.

Hematopoietic: WBC at least 3,000, Platelets at least 75,000.

Hepatic: Not specified.

Renal: Not specified.

Other:

No pregnant women.

Negative pregnancy test required of fertile women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 1989-12; Study Completion 2000-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Waldmann TA, Goldman CK, Bongiovanni KF, Sharrow SO, Davey MP, Cease KB, Greenberg SJ, Longo DL. Therapy of patients with human T-cell lymphotrophic virus I-induced adult T-cell leukemia with anti-Tac, a monoclonal antibody to the receptor for interleukin-2. Blood. 1988 Nov;72(5):1805-16. PMID 2846094
- [Background] Kozak RW, Raubitschek A, Mirzadeh S, Brechbiel MW, Junghans RP, Gansow OA, Waldmann TA. Nature of the bifunctional chelating agent used for radioimmunotherapy with yttrium-90 monoclonal antibodies: critical factors in determining in vivo survival and organ toxicity. Cancer Res. 1989 May 15;49(10):2639-44. PMID 2785435